CLINICAL TRIAL: NCT01685593
Title: A Controlled Randomized Trial Examining the Ability of the Mott Compression Bonder to Decrease Postoperative Pain in Gynecologic Abdominal Laparotomy Patients.
Brief Title: Abdominal Binder Study to Decrease Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edward R. Kost, M.D., Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C.2001.128
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Postoperative Pain
Keywords: abdominal binder
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- regular bandage (Sham Comparator): no abdominal binder
  Interventions: Other: no binder
- abdominal binder (Experimental): binder
  Interventions: Device: abdominal binder

INTERVENTIONS:
Device: abdominal binder
  Arms: abdominal binder
Other: no binder
  Arms: regular bandage

SUMMARY:
We conducted a controlled randomized trial examining the ability of the Mott abdominal Compression Binder to decrease postoperative pain in gynecologic abdominal laparotomy patients

ELIGIBILITY:
Inclusion Criteria:

* gynecologic abdominal laparotomy patients

Exclusion Criteria:

* non gynecologic abdominal laparotomy patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2001-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 24 hours
  linear pain scale

SECONDARY OUTCOMES:
ambulations in 24 hours postoperatively | 24 hours
  number ambulations

OTHER OUTCOMES:
amount morphine used in 24 hours postoperatively | 24 hours
  mg morphine

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States